CLINICAL TRIAL: NCT02208986
Title: GnRHa Trigger in Asian Oocyte Donors Co-treated With a GnRH Antagonist - a Dose Finding Study
Brief Title: GnRHa Trigger in Asian Oocyte Donors- a Dose Finding Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); The Fertility Clinic, Skive Regional Hospital, Denmark (Unknown); Aarhus University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_01_2014
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Normal Oocyte Donors
Keywords: GnRH antagonist; GnRH agonist trigger; Oocyte donor
MeSH Terms: interventions — Triptorelin Pamoate; Powders; Solvents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.2mg Triptorelin (Active Comparator): Ovulation trigger with 0.2mg Triptorelin in one subcutaneous injection.
  Interventions: Drug: Triptorelin
- 0.3mg Triptorelin (Active Comparator): Ovulation trigger with 0.3mg Triptorelin in one subcutaneous injection.
  Interventions: Drug: Triptorelin
- Active Comparator: 0.4mg Triptorelin (Active Comparator): Ovulation trigger with 0.4mg Triptorelin in one subcutaneous injection.
  Interventions: Drug: Triptorelin

INTERVENTIONS:
Drug: Triptorelin — Triptorelin is given by s.c injection for ovulation triggering.
  Other Names: Diphereline 0.1 mg powder and solvent

SUMMARY:
The aim of this randomized single center study is to explore the most optimal dose of GnRHa used for triggering of final oocyte maturation in IVF. The study group will consist of oocyte donors who have GnRHa trigger as a standard trigger concept.

Hypothesis: In an Asian oocyte donor population, the use of 0.2 mg, 0.3mg or 0.4 mg of GnRHa will lead to the retrieval of comparable numbers of mature oocytes (MII) and good quality embryos. Moreover, the reproductive outcome in the recipients will be similar regardless of the dose of GnRHa used for trigger.

DETAILED DESCRIPTION:
Methods

A randomized controlled single center study. All oocyte donors, fulfilling the inclusion criteria, will be eligible for inclusion after randomization.

Stimulation, monitoring, oocyte pick-up in donors and embryo transfer in recipients On day two of the cycle, - i.e. prior to commencing stimulation with long acting FSH (Elonva) - donors will be randomized to one of three groups, using different doses of GnRHa (Triptorelin) for trigger. Stimulation will be performed according to the standard stimulation protocol of the clinic, using Elonva followed by co-treatment with a GnRH antagonist from day 5 of stimulation . The dose of Elonva used for stimulation will be either 100 or 150 µg according to the weight of the patient. The first transvaginal ultrasound scan (TVUS) will be performed after seven or eight days after the Elonva depot injection. As soon as two follicles have reached a size of ≥ 17mm, triggering of final oocyte maturation will be performed with one single bolus of Triptorelin, 0.2 mg, 0.3mg or 0.4 mg. The timing of the trigger will be 6 AM for all groups and the oocyte pick-up (OPU) will be performed after 34 hours, according to the usual practice of the clinic. Importantly, each patient will be asked to check the presence of an LH surge via a urine LH detection kit at 4 hours after the trigger bolus has been administered. Embryo transfer will be performed on day two in all recipients.

Study group I Stimulation according to the abovementioned and ovulation trigger with 0.2mg Triptorelin. All other procedures will be performed according to the practice of the clinic.

Study group II Stimulation according to the abovementioned and ovulation trigger with 0.3mg Triptorelin. All other procedures will be performed according to the practice of the clinic.

Study group III Stimulation according to the abovementioned and ovulation trigger with 0.4mg Triptorelin. All other procedures will be performed according to the practice of the clinic.

Randomization Randomization will be performed using sealed envelopes developed via a computer generated list with blocks of twelve. The randomization will be performed on day two of the cycle. Doctors will be blinded to the randomization, but not patients and nurses.

Follicular fluid (FF) collection FF from the first punctured follicle on each side will be collected and cryo-preserved at -20 degrees for subsequent analysis of steroids.

Granulosa cell gene-expression analysis Cumulus and mural granulosa cells will be preserved and snap-frozen from a sub-group of 10 patients in each group. The primary subsequent analysis will focus on possible differences in LHR gene expression according to GnRHa trigger dose.

ELIGIBILITY:
Inclusion Criteria:

Oocyte donors who meet the following criteria:

* Age 18 - 35
* BMI < 28kg/m2
* Normal ovarian reserve, defined by AMH > 1.25 ng/ml or AFC ≥ 6 measured within two months prior to stimulation start
* Receiving GnRH-antagonist protocol for ovarian stimulation,
* Agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
* Have given written informed consent with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Previous poor response (≤ 3 oocytes) after high dose FSH stimulation
* Chronical medical conditions like Diabetes, Crohns disease, Thyroid disease, Hepatitis B and Sexually Transmitted Diseases Simultaneous participation in an interventional clinical trial.
* Concommitant use of either LH or hMG/uFSH preparations in study cycle

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes | 30 minutes after oocyte retrieval completed

SECONDARY OUTCOMES:
Day of bleeding after oocyte pick-up | in 2 weeks after oocyte pick-up
Clinical pregnancy | 5 weeks after oocyte pick-up

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — CGRH, School of Medicine, Vietnam National University HCMC, Vietnam; Lan TN Vuong, MD, Principal Investigator — Department of Obstetrics and Gynecology, University of Medicine and Pharmacy HCMC, Ho Chi Minh City, Vietnam; Peter Humaidan, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- My Duc Hospital, IVFMD, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong TN, Ho MT, Ha TD, Phung HT, Huynh GB, Humaidan P. Gonadotropin-releasing hormone agonist trigger in oocyte donors co-treated with a gonadotropin-releasing hormone antagonist: a dose-finding study. Fertil Steril. 2016 Feb;105(2):356-63. doi: 10.1016/j.fertnstert.2015.10.014. Epub 2015 Oct 31. PMID 26523330